CLINICAL TRIAL: NCT04592679
Title: FES Cycling Cost-Effectiveness Analysis in Rehabilitation for Persons Affected by Complete Spinal Cord Injury, an Experience From Two Italian Hospitals
Brief Title: Cost-Effectiveness Analysis of a Rehabilitation Protocol With FES Cycling in Persons With Complete SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Matteo Olivieri, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3879B
Record Dates: First submitted 2020-09-28; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: FESD; Rehabilitation; Spinal Cord Injuries; Complete Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES-C (Experimental)
  Interventions: Device: FES-C
- Standard (Active Comparator)
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Device: FES-C — The participants were submitted to 20 sessions of FES-C three/five times per week. Each session lasted about 30'.
  Arms: FES-C
Other: Standard Treatment — The participants were submitted to 20 sessions of standard rehabilitation for lower limbs with manual mobilization, three/five times per week. Each session lasted about 30'.
  Arms: Standard

SUMMARY:
20 patients were recruited by two hospitals (AOUP and AOUC) in Italy from January 2015 to January 2018. The participants have been addressed to two different groups: the ones recruited by the AOUP were submitted to an experimental protocol of rehabilitation with FES Cycling, the ones recruited by the AOUC were submitted to a standard protocol of manual mobilization.

The primary outcome was the thigh circumferences measured at 4 different levels (5-10-15-20 cm) from the superior margin of the patella, while the secondary outcomes were the muscle tone evaluated with Modified Ashworth Scale (MAS) and the sensation of pain registered with International Spinal Cord Injury - Pain Basic Data Set (ISCI-P).

From these outcomes the Quality Adjusted Life Years (QALYs) was obtained. The costs of the two treatments were calculated through a consultation process with the Competent Offices of the two hospitals. The QALYs and the costs were used to calculate the Incremental Cost-Effectiveness Ratio (ICER) in order to verify the cost-effectiveness ratio of the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* complete spinal cord injury
* loss of gait function
* any episode of autonomic dysreflexia
* any important range of motion limitation to hips, knees or ankles
* eccitability of the muscles
* FES tollerability

Exclusion Criteria:

* cognitive deficits
* psychiatric diseases
* cancer
* recent fractures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Incremental Cost-Effectiveness Ratio | 3 years
  QALYs/costs of the two treatments, the ICER could variate from -100'000 to 100'000 QALYs/€
Thigh Circumferences | 3 years
  The primary outcome was the thigh circumferences measured at 4 different levels (5-10-15-20 cm) from the superior margin of the patella, the raging of the improvement could be from 0 to 50 cm

SECONDARY OUTCOMES:
Quality Adjusted Life Years (QALYs) | 3 years
  It consists in the use of a scale 0 (death) - 1 (the best possible state of health) for the improvements of the patients
Costs | 3 years
  the costs of the two treatments could variate from 0 to 50'000 €
Muscle tone | 3 years
  Muscle tone evaluated with "Modified Ashworth Scale" (MAS), 0-5 points, an higher result means more spasticity
Sensation of pain | 3 years
  Sensation of pain evaluated with "International Spinal Cord Injury - Pain Basic Data Set" 0-30 points, an higher result means more sensation of pain (ISCI-P).

IPD SHARING:
Plan to Share IPD: Undecided